CLINICAL TRIAL: NCT06315569
Title: The Effect of Exercise at Different Time Intervals on Hyperuricemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20242030-C-1
Record Dates: First submitted 2024-02-18; First posted 2024-03-18 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (two 3000m runs 24 hours apart) (Experimental): Run a second 3000m run 24 hours after completing the first 3000m run
  Interventions: Behavioral: Run 3000 meters
- Group B (two 3000m runs 48 hours apart) (Experimental): Run a second 3000m run 48 hours after completing the first 3000m run
  Interventions: Behavioral: Run 3000 meters

INTERVENTIONS:
Behavioral: Run 3000 meters — Participants in both groups were asked to do two 3,000-meter runs at different intervals

SUMMARY:
The study aim is to explore the correlation between exercise and hyperuricemia, find out the metabolic rule of uric acid after exercise, and provide scientific evidence and clinical guidance for how to exercise scientifically and reasonably in patients with hyperuricemia. This trial is a multicenter, prospective, randomized controlled clinical trial with 100 participants. Inclusion criteria: 1. Patients with hyperuricemia (fasting uric acid > 420μmol/L twice on different days); 2. Men aged between 18 and 35; 3. Able to complete baseline fitness test (3000m run time less than 14 minutes); 4. Fully informed consent, signed informed consent exclusion criteria: 1. Patients with heart, liver and kidney insufficiency. 2. Subjects suffering from severe or uncontrollable organic diseases may interfere with study parameters such as hypertension, hyperlipidemia, hyperglycemia, tumor, cardiovascular, lung and digestive diseases. 3. Patients with secondary hyperuricemia caused by other diseases. 4. Take any drugs that may cause uric acid changes in the past 4 weeks. 5. Those who have related motor function or other factors are easy to cause discomfort after exercise. 6. Those who have mental illness or communicate do not cooperate during the test.

A total of 100 participants participated in the study（Group A n = 50 ; Group B n = 50 ）. The subjects are divided into two groups, designated as A and B. Following the completion of the grouping, all subjects complete the initial 3000 m run. The second 3000 m run is performed on the seventh day following the initial run. The interval between the third run and the second run in Group A is 24 hours, while the interval in Group B is 48 hours. During the 48-hour observation period after each exercise, the changes of uric acid after exercise were explored. To provide scientific evidence and clinical guidance for patients with hyperuricemia how to exercise scientifically and rationally.

Patients must meet all inclusion and exclusion criteria to be eligible to participate in the study. After determining patients' eligibility for the study, the researcher should fully explain the nature, purpose, risks and benefits of the study to the subjects before the study, and assure the patients that they have the right to withdraw at any time after agreeing to participate in the study, and the subjects should sign a written informed consent after fully considering and agreeing to participate in the study. The process of obtaining informed consent should be correctly recorded in all case report forms in this study.

Baseline data such as blood uric acid, blood biochemistry, blood routine, urine routine, uric acid, and demographic characteristics were collected after the patients were enrolled.

The patients were randomly divided into two groups: Group A and Group B. Within 48 hours after each 3000m exercise, the subjects' blood uric acid was detected after exercise 1 hour, 2 hours, 3 hours, 12 hours, 24 hours, 36 hours, 48 hours.

From January 2024 to February 2024, we plan to draft clinical study protocols, investigator manuals, case reports, informed consent forms and other documents, and submit them to the Ethics Committee of the research sponsor for review and approval; February 2024 - March 2024: Complete the training of all researchers and officially start the research; March 2024 - August 2024: Participants were enrolled for the experiment; August 2024 - November 2024: collate and collect data, conduct statistical analysis, and confirm research results

ELIGIBILITY:
Inclusion Criteria:

* Patients with hyperuricemia (fasting uric acid > 420μmol/L twice on different days);
* Men aged between 18 and 35;
* Able to complete baseline fitness test (3000m run time less than 14 minutes);
* Fully informed consent, sign informed consent.

Exclusion Criteria:

* Patients with heart, liver and kidney insufficiency;
* Subjects suffering from severe or uncontrollable organic diseases may interfere with study parameters such as hypertension, hyperlipidemia, hyperglycemia, tumor, cardiovascular, lung and digestive diseases;
* Patients with secondary hyperuricemia caused by other diseases;
* Take any drugs that may cause uric acid changes in the past 4 weeks;
* Those who have related motor function or other factors are easy to cause discomfort after exercise；
* Those who have mental illness or communicate do not cooperate during the test.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Uric acid metabolism in patients with hyperuricemia after exercise | 1 week
  Monitoring changes in uric acid levels after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi’an, Shanxi, China